CLINICAL TRIAL: NCT07010757
Title: Testing an Integrated PTSD and Weight Management Intervention: A Hybrid Type 1 Trial
Acronym: HARPP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 24-046; HX003961-01A1 (Other Grant/Funding Number: U.S. Department of Veterans Affairs)
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: PTSD; Obesity
Keywords: Veteran; behavioral weight management; cognitive processing therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Obesity

STUDY DESIGN:
Intervention Model Description: Testing an integrated treatment that combines PTSD and weight management care, using behavioral and pharmacologic approaches, relative to usual care in a randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Staff will not be able to predict treatment assignment at the point of randomization. Assessors, and biostatisticians will be masked until after 12-month data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): Participants in the control condition will receive the following:
  1. Referral to MOVE!; they will select a MOVE! that fits their schedule (at VAPS MOVE! is a 12-week group).
  2. Standard CPT in 60-minute individual sessions, delivered by 4 CPT-trained psychotherapists (different therapists than intervention arm therapists to avoid contamination).
  3. One non-visit consult medication review using the same procedures and template outlined above. After the non-visit consult, the Dr. will alert the Veteran's relevant usual care team member(s) via the non-visit consult template in the medical record. They will not have direct contact with control participants, but the study team will monitor for safety following any medication changes.
  Interventions: Behavioral: control arm for HARPP trial
- intervention (HARPP) (Experimental): In HARPP, MOVE! and CPT are delivered in up to 16 individual psychotherapy sessions. While all CPT content is included, it is slightly tailored to address factors that interfere with health behavior change (e.g., hypervigilance that hinders community-based physical activity). All MOVE! materials are included; MOVE! uses cognitive-behavioral techniques and autonomy-supporting counseling to promote physical activity and healthy eating. HARPP targets other PTSD-related barriers to recovery and healthy lifestyles by promoting sleep and relationship quality, and community engagement. HARPP participants receive at least one medication management consultation (review by clinician and telephone session) focused on currently may cause weight gain and AOM options. When relevant and based upon Veteran interest, medications are changed or prescribed, in coordination with the Veteran's psychiatric and primary care teams.
  Interventions: Behavioral: HARPP

INTERVENTIONS:
Behavioral: HARPP — In HARPP, MOVE! and CPT are delivered in up to 16 individual psychotherapy sessions. While all CPT content is included, it is slightly tailored to address factors that interfere with health behavior change (e.g., hypervigilance that hinders community-based physical activity). All MOVE! materials are included; MOVE! uses cognitive-behavioral techniques and autonomy-supporting counseling to promote physical activity and healthy eating. HARPP targets other PTSD-related barriers to recovery and healthy lifestyles by promoting sleep and relationship quality, and community engagement. HARPP participants receive at least one medication management consultation (review by clinician and telephone session) focused on currently may cause weight gain and AOM options. When relevant and based upon Veteran interest, medications are changed or prescribed, in coordination with the Veteran's psychiatric and primary care teams.
  Arms: intervention (HARPP)
Behavioral: control arm for HARPP trial — Participants in the control condition will receive the following:
  1. Referral to MOVE!; they will select a MOVE! that fits their schedule (at VAPS MOVE! is a 12-week group).
  2. Standard CPT in 60-minute individual sessions, delivered by 4 CPT-trained psychotherapists (different therapists than intervention arm therapists to avoid contamination).
  3. One non-visit consult medication review using the same procedures and template outlined above. After the non-visit consult, the Dr. will alert the Veteran's relevant usual care team member(s) via the non-visit consult template in the medical record. They will not have direct contact with control participants, but the study team will monitor for safety following any medication changes.
  Arms: control group

SUMMARY:
Obesity and post-traumatic stress disorder (PTSD) are common among Veterans. PTSD increases risk for obesity, impacting functioning, health, quality of life, and premature mortality. Use of proven treatments for PTSD and obesity in VA is low. Furthermore, Veterans with PTSD lose less weight than those without PTSD in VA's national weight management program. Based on pilot work, an integrated treatment that combines PTSD and weight management care-using behavioral and pharmacologic approaches-may improve weight and PTSD. Whether it improves these outcomes more than standard VA care is unknown, which is the focus of this study. The study also seeks to understand factors that would interfere with and facilitate implementing the program in VA if it is effective. This Veteran-centered program may be a more efficient and effective treatment for Veterans with PTSD and obesity, addressing both physical and mental health.

DETAILED DESCRIPTION:
Background: Obesity and post-traumatic stress disorder (PTSD) are highly prevalent among Veterans. PTSD increases risk for obesity and related conditions, in part due to PTSD symptoms interfering with physical activity and healthy diet. VA offers effective evidence-based behavioral and pharmacologic weight management and PTSD treatments, but utilization is low. Veterans with PTSD also lose less weight than those without mental health conditions in VA's MOVE! behavioral weight management program. In response, the investigators developed HARPP-an integrated weight and PTSD treatment-to promote improved access, efficiency, and outcomes. HARPP is a manualized 16-session individually-delivered treatment that combines VA's MOVE! behavioral weight management program and cognitive processing therapy (CPT), enhanced to address obesity-PTSD intersections, and medication review and management. The latter focuses on identifying obesogenic medications that could be changed and eligibility for anti-obesity medications (AOM) through chart review, ~2-3 virtual visits with an obesity specialist, and close coordination with Veterans' care teams. In a pilot of HARPP among 7 Veterans, participants reported high satisfaction, and experienced substantial weight loss and PTSD symptom reduction. HARPP effectiveness must be tested in a randomized controlled trial (RCT).

Significance/Impact: The study aligns with VA and HSR priorities, given its focus on meaningful Veteran engagement to develop and test a novel, Veteran-centered, whole health intervention focused on improving access and outcomes for Veterans with PTSD, a priority VA population. This study's identification of implementation determinants would place effectiveness findings in context and facilitate translation to clinical care if HARPP is effective. This study will also yield insights about how weight management and PTSD care can be enhanced broadly. For example, the medication protocol and templates could be of use broadly in VA.

Innovation: HARPP is the first integrated treatment designed to address obesity and PTSD simultaneously.

Specific Aims: The investigators will randomize 182 Veterans with PTSD and obesity to control (standard CPT, referral to standard MOVE!, and one non-visit consult medication review) or intervention (HARPP, described above) to address the following aims: 1) Test whether intervention participants have greater absolute weight loss in pounds and PTSD symptom reduction relative to controls at 6 (secondary outcomes) and 12 months (co-primary outcomes); 2) Assess whether taking AOM mediates the relationship between HARPP and 12-month weight loss; and 3) Assess implementation determinants (acceptability, feasibility, fidelity, and cost).

Methodology: The investigators propose to conduct a hybrid type 1 RCT among Veterans with PTSD and obesity to test the primary hypothesis that HARPP participants will have greater 12-month absolute weight loss in pounds and PTSD symptom reduction relative to Veterans enrolled in the control group. The Veteran Engagement Group will consult throughout the study, ensuring Veteran-centeredness.

Next Steps/Implementation: If trial findings suggest HARPP is effective, the study team will partner with Veterans and operational leaders to develop a HARPP implementation package that will be tested in a multi-site hybrid type 2 trial, findings of which will inform broad VA implementation. Implementation activities would be coordinated with existing local, VISN, and national operational partners. If HARPP is not effective, Aims 2 and 3 will help understand how Veterans with PTSD and obesity could be better supported in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Current PTSD Diagnosis per Clinician-Administered PTSD Scale for DSM-5 (CAPS)
2. Obesity: BMI of 30 kg/m2
3. Enrolled in VAPS primary care to ensure safety and facilitate HARPP's medication component
4. Willing to do intervention or control and assessments

Exclusion Criteria:

1. Not fluent in English, severe hearing loss, no phone access
2. Recent MOVE! or CPT participation (2 visits in past 2 months)
3. Had bariatric surgery in past 6 months or plans to receive it in next 12 months
4. At least 1 fill of AOM in the past 90 days
5. Current pregnancy
6. Any history of a bulimia diagnosis and/or meets criteria for bulimia
7. Cannot participate due to a) acute substance use, mental health, or medical exacerbation or b) at least moderate neurologic conditions, e.g., dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
12-month absolute weight change in pounds | 12 months post-baseline
  Body weight will be measured on a study scale at baseline and 12 months following baseline. This study's co-primary aim is to test whether intervention participants have greater 12-month weight loss, relative to controls.
12-month absolute PTSD symptom severity change | 12 months post-baseline
  PTSD symptom severity will be measured via self-report on the PTSD Checklist for DSM-5 at baseline and 12 months following baseline. This study's co-primary aim is to test whether intervention participants have greater 12-month PTSD symptom reduction, relative to controls.

SECONDARY OUTCOMES:
6-month absolute weight change in pounds | 6 months post-baseline
  Body weight change from baseline to 6 months (measured by assessing weight on a study scale at baseline and 6 months following baseline) will be compared between intervention and control groups.
6-month absolute PTSD symptom severity change (PCL-5) | 6 months post-baseline
  PTSD symptom severity will be measured via self-report on the PTSD Checklist for DSM-5 at baseline and 6 months following baseline. Symptom severity change from baseline to 6 months will be compared between intervention and control groups.
6-month absolute PTSD symptom severity change (CAPS-5-R) | 6 months post-baseline
  PTSD symptom severity will be measured via a clinician-administered measure, the CAPS-5-R as a secondary outcome: change in absolute PTSD symptom severity at 6 months as measured with the CAPS-5.

OTHER OUTCOMES:
12-month anti-obesity medication prescription | 12 months post-baseline
  Whether or not (yes vs. no) participant had at least 1 pharmacy fill of Anti-obesity medication in the 12 months post-baseline, per VA pharmacy data. Will be assessed as a mediator in an exploratory analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine D Hoerster, PhD MPH BA, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No